CLINICAL TRIAL: NCT02251171
Title: A Single-centre Open-label Study in Healthy Adult Volunteers to Determine the Effects of Steady-state TPV/RTV (500 mg/200 mg) on the Single-dose Pharmacokinetics of Rifabutin (MYCOBUTIN®) 150 mg, and the Effects of Single-dose Rifabutin (150 mg) on the Steady-state Pharmacokinetics of TPV 500 mg (Co-administered With RTV 200 mg)
Brief Title: Effects of Steady-state TPV/RTV on the Single-dose Pharmacokinetics of Rifabutin and the Effects of Single-dose Rifabutin on the Steady-state Pharmacokinetics of TPV in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.44
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Rifabutin

ARMS (1):
- TPV/RTV - Rifabutin (Experimental): Day 1: single dose Rifabutin
  Days 8-20: morning and evening doses of Tipranavir/Ritonavir
  Day 15: single dose Rifabutin
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Rifabutin

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
  Other Names: Norvir-SEC®
Drug: Rifabutin
  Other Names: Mycobutin®

SUMMARY:
Study to determine the effects of steady-state Tipranavir (TPV) / Ritonavir (RTV) (500mg/200mg bid) on the single-dose pharmacokinetics of Rifabutin (RFB) and to determine the effects of single-dose RFB on the steady-state pharmacokinetics of TPV 500mg (co-administered with RTV 200mg)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 60 years of age inclusive
2. A Body Mass Index (BMI) between 18 and 29 kg/m2
3. Signed informed consent prior to trial participation
4. Ability to swallow multiple large capsules without difficulty
5. Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity was less than or equal to Grade 1, based on the AIDS Clinical Trials Group (ACTG) Grading Scale. All abnormal laboratory values greater than Grade 1 are subject to approval by the trial clinical monitor
6. Acceptable medical history, physical examination, and 12-lead ECG are required prior to entering the treatment phase of the study. The requirement for chest X-ray is left to the investigator's discretion
7. Willingness to abstain from the following starting 14 days prior to any administration of study drug up until the end of the study:

   * Grapefruit or grapefruit juice
   * Red wine
   * Seville oranges
   * St. John's Wort or Milk Thistle
8. Willingness to abstain from alcohol starting 2 days prior to administration of any study drug up to the end of the study
9. Willingness to abstain from the following within 72 hours of pharmacokinetic (PK) sampling:

   * Garlic supplements
   * Methylxanthine containing drinks (coffee, tea, cola, energy drinks, chocolate, etc.)
10. Willingness to abstain from over the counter herbal medications for the duration of the study
11. Have been non-smokers for 3 months
12. Willingness to abstain from vigorous physical exercise during intensive PK study Days 1, 14, and 15
13. Reasonable probability for completion of the study

Exclusion Criteria:

As a guideline, subjects who have abnormal laboratory values at screening, and who are taking prescription medications are excluded:

1. Female subjects with reproductive potential who:

   * Have positive serum β-human chorionic gonadotropin at Visit 1, or on study Day 0 or study Day 1
   * Have not been using a barrier contraceptive method for at least 3 months prior to Visit 3 (study Day 1)
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during the trial and 60 days after completion/termination
   * Are breast-feeding
2. Participation in another trial with an investigational medicine within 60 days prior to study Day 0 (Visit 2)
3. Use of any medication listed in Protocol within 30 days prior to study Day 0 (Visit 2)
4. Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to study Day 0 and for the duration of the study. Use of Depo-Provera is excluded for six months prior to study Day 0
5. Use of hormone replacement therapy within 1 month prior to study Day 0 and for the duration of the study
6. Administration of antibiotics within 10 days prior to study Day 0 (Visit 2) or during the trial
7. History of acute illness within sixty (60) days of study Day 0. Subjects are excluded if they have an acute illness greater than sixty days prior to study Day 0 if, in the opinion of the investigator, the subject did not qualify as a healthy volunteer
8. History of thrombotic disease
9. History of migraine headache
10. Have serological evidence of hepatitis B or C virus
11. Have serological evidence of exposure to HIV
12. Recent history of alcohol or substance abuse (within 1 year of screening)
13. Blood or plasma donations within 30 days prior to study Day 0 (Visit 2) or during the trial
14. Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min. For subjects with a resting heart rate below 50, or above 90, the investigator may discuss their exclusion with the clinical monitor on a case-by-case basis
15. Subjects with history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV, RTV or RFB to the subject
16. Subjects who have taken (within 7 days prior to study Day 0) or are taking any over-the-counter or prescription drug that, in the opinion of the investigator in consultation with the clinical monitor, might interfere with either the absorption, distribution or metabolism of the test substances
17. Known hypersensitivity to TPV, RTV, RFB, or sulphonamide class of drugs
18. Inability to adhere to the protocol
19. Cautions or warnings in the RTV and RFB package insert which, in the judgment of the investigator, should exclude a subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-08; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of the analytes in plasma (Cmax) | up to 144 hours after drug administration
Drug concentration of the analytes in plasma at 12 hours after administration (Cp12h) | up to 12 hours after drug administration
Area under plasma concentration time curve from 0-12 hours (AUC0-12h) | up to 12 hours after drug administration
Area under the plasma drug concentration-time curve from time zero to infinity of the analytes (AUC0-∞) | up to 144 hours after drug administration

SECONDARY OUTCOMES:
Oral clearance (CL/F) | up to 144 hours after drug administration
Time of maximum concentration (Tmax) | up to 144 hours after drug administration
Volume of distribution (V) | up to 144 hours after drug administration
Apparent terminal half life (t1/2) | up to 144 hours after drug administration
Number of subjects with adverse events | up to 24 days
Number of subjects with abnormal changes in laboratory parameters | up to 21 days